CLINICAL TRIAL: NCT03892239
Title: The Effectiveness of a Running-related Injury Prevention Program in Brazilian Runners: a Randomised Controlled Trial
Brief Title: The Effectiveness of a Running-related Injury Prevention Program in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Luiz Carlos Hespanhol Junior, Associate Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UNICID 20
Record Dates: First submitted 2019-02-05; First posted 2019-03-27 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Running-related Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Monitoring and suggestion of training progress. Behaviour change strategy based on increasing knowledge.
  Interventions: Behavioral: RunIn3 Prevention Program
- Control (Active Comparator): Monitoring and suggestion of training progress.
  Interventions: Behavioral: Feedback Based Surveillance

INTERVENTIONS:
Behavioral: RunIn3 Prevention Program — The intervention will be delivered online. Every two weeks we will send a link to participants that will direct them to an online questionnaire. The online questionnaire will collect information on complaints and symptoms related to running, and the volume, intensity and frequency of running practice within the 2-week period. If the participant reports any symptom and if she/he accepts a suggestion regarding running training, an algorithm embedded in the online system will automatically suggest a training volume for the next two weeks based on the distance and/or duration reported by the participant.
  Through a website we will make available informative texts, videos and infographics in order to increase the participant's knowledge regarding topics such as: musculoskeletal symptoms; foot strike patterns; training workload; running shoes; warming-up/cooling-down, stretching; and concomitant strength training.
  Arms: Intervention
Behavioral: Feedback Based Surveillance — The intervention will be delivered online. Every two weeks we will send a link to participants that will direct them to an online questionnaire. The online questionnaire will collect information on complaints and symptoms related to running, and the volume, intensity and frequency of running practice within the 2-week period. If the participant reports any symptom and if she/he accepts a suggestion regarding running training, an algorithm embedded in the online system will automatically suggest a training volume for the next two weeks based on the distance and/or duration reported by the participant.
  Arms: Control

SUMMARY:
Running is effective in increasing levels of physical activity and promotes a number of beneficial health effects. However, running can lead to running- related injuries (RRI). In theory, such injuries can be avoided with the implementation of prevention programs. But in practice, there is a paucity of prevention programs that are effective in reducing the risk of RRIs. In a previous study, the investigators developed an RRI prevention program using the Intervention Mapping framework. The RRI prevention program was named RunIn3. The present study will evaluate the effectiveness of the RunIn3 RRI prevention program.

Objective: To investigate the effectiveness of an RRI prevention program (i.e., RunIn3).

There will be recruited 530 runners of the state of São Paulo aged 18 years or older. After inclusion, participants will be randomly assigned and allocated in two groups: (1) intervention group, which will be the target of the implementation of the RunIn3 prevention program; and (2) control group, which will receive a minimal intervention (i.e., feedback based on surveillance).

ELIGIBILITY:
* Running experience of at least three months;
* Residents of the state of São Paulo;
* No running-related injury (RRI) at baseline;
* No history of RRI in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Running-related injuries (RRI) | After 12 months from baseline
  Symptoms and complaints related to running will be measured and monitored by the Brazilian-Portuguese version of the Oslo Sports Trauma Research Center (OSTRC) Questionnaire on Health Problems (OSTRC-Br).

SECONDARY OUTCOMES:
Behaviour | After 12 months from baseline
  The preventive behaviours towards running-related injuries (RRI) adopted or modified will be collected using an online questionnaire that will be composed of questions with 7-point Likert scales (-3 to +3).
Costs | After 12 months from baseline
  The cost data will be collected through a questionnaire composed of open-ended and multiple choice questions regarding direct costs (medical and non-medical costs) and indirect costs (work absenteeism) regarding participants' health related to running practice.
Incremental cost-effectiveness ratio (ICER) | After 12 months from baseline
  The incremental cost-effectiveness ratio (ICER) will be estimated taking total costs and the effects on running-related injuries (RRI).

CONTACTS AND LOCATIONS:
Overall Officials: Caio S Vallio, PT, Principal Investigator — Universidade Cidade de São Paulo (UNICID); Luiz Hespanhol, PhD, Study Chair — Universidade Cidade de São Paulo (UNICID)
Locations (1):
- Universidade Cidade de São Paulo (UNICID), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barros PM, Vallio CS, Oliveira GM, Miyamoto GC, Hespanhol L. Cost-effectiveness and implementation process of a running-related injury prevention program (RunIn3): Protocol of a randomized controlled trial. Contemp Clin Trials Commun. 2021 Jan 20;21:100726. doi: 10.1016/j.conctc.2021.100726. eCollection 2021 Mar. PMID 33553800